CLINICAL TRIAL: NCT03358628
Title: Patient-derived Xenograft (PDX) Modeling to Test Drug Response for High-grade Osterosarcoma
Brief Title: Patient-derived Xenograft (PDX) Modeling to Test Drug Response for High-grade Osteosarcoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, GUO WEI, Chief of Musculoskeltal Tumor Center, Peking University People's Hospital
Other Study IDs: 2017PHB278-01
Record Dates: First submitted 2017-11-25; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma; Patient-derived xenograft
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, formalin fixed paraffin embedded blocks, or fresh tumor tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteosarcoma: Osteosarcoma patients with metastatic relapsed or unresectable progressive disease (total n= up to 20) following resection of the primary lesion and adjuvant chemotherapy.
  Interventions: Other: Molecular Profiling & In Vivo drug testing in PDX

INTERVENTIONS:
Other: Molecular Profiling & In Vivo drug testing in PDX — Molecular profiling of host tumour sample and PDX will be performed and analyzed by an expert panel. In vitro drug testing using organoid culture generation may also be performed if sufficient fresh tissue is available. Matched treatment recommendation based on profiling and in vivo PDX drug testing results will be made, if available.

SUMMARY:
By obtaining clinical specimens from participants with high-grade bone and soft tissue sarcomas to establish and profile as freshly implanted tumors in mice, the aim of this study is to identify agents with predicted activity in the host patient while also potentially providing them with individualized cancer treatment options

DETAILED DESCRIPTION:
Patient-derived xenografts (PDX) are increasingly used as tools for drug development in pre-clinical settings, and have been shown to recapitulate the histology and behavior of the cancers from which they are derived. Although, they have been commonly used productively as pre-clinical disease models to study disease biology and drug response, they have not been used prospectively to inform clinical management. PDX have been employed to inform clinical decision-making in small studies, which have shown high concordance between individual PDX and patient responses to therapy. While encouraging, the role of this approach in bone and soft tissue sarcomas and in the context of genomic drug matching strategies remains undefined. This has created an opportunity to evaluate the utility of PDX as clinical predictors to direct the use of chemo- and targeted therapies in combination with comprehensive genomic and epigenetic analysis for patients with bone and soft tissue sarcomas.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years;
2. Diagnosis confirmed histologically and reviewed centrally;
3. Prior treatment (completed >4 weeks before trial entry) consisted of standard high-grade osteosarcoma chemotherapy agents including doxorubicin, cisplatin, high-dose methotrexate, and ifosfamide; metastatic relapsed and unresectable progressive disease (PD);
4. Eastern Cooperative Oncology Group performance status 0-1 with a life expectancy >3 months;
5. Adequate renal, hepatic, and hemopoietic function;
6. Normal or controlled blood pressure;
7. Surgery and/or radiotherapy completion at least 1 month before enrollment.

Exclusion Criteria:

1. Central nervous system metastasis;
2. Have had other kinds of malignant tumors at the same time;
3. Cardiac insufficiency or arrhythmia;
4. Uncontrolled complications, such as diabetes mellitus and so on;
5. Coagulation disorders;
6. Urine protein≥ ++;
7. Pleural or peritoneal effusion that needs to be handled by surgical treatment;
8. Combined with other infections or wounds.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-grade osteosarcoma referred to, or being treated at Peking University People's Hostpital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2020-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Measure of drug sensitive PDX to a panel of drugs as a predictor of clinical response in matched host | up to 2 years
  Sensitivity measured by tumor growth inhibition (>80%) or objective tumor response (regression) as per Response Evaluation Criteria In Solid Tumors (RECIST) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, MD, PhD, Principal Investigator — Peking University People's Hospital